CLINICAL TRIAL: NCT06907277
Title: Dexmedetomidine-based Enhanced Recovery After Cardiac Surgery Improves Outcome Regarding Analgesia, Sleep Disorders, and Postoperative Delirium
Brief Title: Dexmedetomidine Enhancing the Recovery After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohammed Abd ElRahman Hammed, Assistant Lecturer of Anesthesia, Pain & ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC 17-11-2024
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Post-cardiac Surgery
MeSH Terms: interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: Lidocain
- Group F (Active Comparator)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine (DXM) loading dose of 0.6 µg/kg followed by DXM infusion given at a rate of 0.4 ml/kg/h and was provided as 0.15 µg/kg/h for 24-h PO.
  Arms: Group D
Drug: Fentanyl — A bolus of fentanyl 5 µg/kg followed by an intraoperative (IO) fentanyl infusion of 3-5 µg/kg/h that was continued as PO analgesia for 24 hours in a dose of 0.3 µg/kg/h.
  Arms: Group F
Drug: Lidocain — Lidocaine (LID) loading dose (1 mg/kg) followed by a continuous infusion till 24 h PO as 1.5 mg/kg/h.
  Arms: Group D

SUMMARY:
Enhanced Recovery After Surgery (ERAS) aims to facilitate a quicker and smoother recovery period following surgical procedures. The implementation of these protocols may lead to patients returning to their daily activities sooner, experiencing greater satisfaction with their care, and potentially encountering fewer complications, ultimately contributing to shorter hospital stays. However, a common challenge in the postoperative phase is postoperative delirium(POD). This complication can lead to both immediate and long-term cognitive impairments, negatively impact overall health outcomes, and increase the financial burden on the healthcare system. Interestingly, dexmedetomidine, known as DXM, is a medication that selectively targets certain receptors in the brain and offers sedative properties with minimal impact on breathing. This characteristic is noteworthy because it may help regulate sleep patterns and support the preservation of cognitive function during the recovery period.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists Classification (ASA) grade II-III;
* Patients who were planned to have Coronary Artery Bypass Graft (CABG);
* Patients were free of exclusion criteria.

Exclusion Criteria:

* Patients with preoperative high risk for getting Post Operative Delirium or sleep disorders,
* Patients with American Society of Anesthesiologists Classification (ASA) grade>III;
* Patients with heart failure, left ventricle ejection fraction of <25%,
* Patients with uncontrolled diabetes mellitus, coagulopathy, or history of uncompensated renal or hepatic diseases

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Significant Enhancement of Post Operative Recovery Levels After Dexmedetomidine Administration in Cardiac Surgery. | 3 months
  Post-operative recovery was measured on 3 levels: Confusion, Sleep Quality, and Delirium.
  The study focused primarily on postoperative delirium through the Delirium Index, a 7-item questionnaire that graded the severity of delirium in patients with or without dementia. These seven items assess disorders of attention, thought, consciousness, orientation, memory, perception, and psychomotor activity. Each item is scored on a 0-3 scale, with zero indicating the absence of disturbance, while 1-3 indicates mild, moderate, and severe disturbance of the assessed function for a total score ranging between 0 and 21, and higher scores indicate higher delirium severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, El Qalyoubia, Egypt